CLINICAL TRIAL: NCT00128908
Title: Sequential HAART in Treatment Resistant HIV-1 Infected Patients
Brief Title: Sequential HIV Therapy in Treatment Resistant HIV-1 Infected Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not recruit
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch AIDS Fund (Unknown)
Responsible Party: Prof. J. Prins, Academic Medical Center, Amsterdam
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05IAT0061; 2004040 - Dutch AIDS Fund
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infections
Keywords: HIV-1; HAART; sequential HAART; resistance; salvage therapy; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous triple-class therapy (Active Comparator): Patients will be treated with a regimen containing antiretroviral agents from 3 different classes
  Interventions: Drug: Standard Continuous Highly Active Antiretroviral Therapy (HAART)
- Alternating therapy (Experimental): Patients will be assigned to weekly alternating dual-class regimen
  Interventions: Drug: Rapidly Cycled HAART

INTERVENTIONS:
Drug: Standard Continuous Highly Active Antiretroviral Therapy (HAART)
  Arms: Continuous triple-class therapy
Drug: Rapidly Cycled HAART
  Arms: Alternating therapy

SUMMARY:
This is an open label, crossover pilot study to explore the safety and efficacy of a rapid cycling regimen of antiretroviral combination therapy in HIV-1 infected patients with virus harboring genotypic resistance to at least three classes of antiretroviral therapy.

DETAILED DESCRIPTION:
Mathematical modeling has suggested that cyclic use of antiretroviral therapy can be an effective strategy in lowering viral load in HIV-1 infected patients when regular triple drug combinations have lost efficacy due to the emergence of HIV resistance mutations.

This is an open label, crossover pilot study to explore the safety and efficacy of a rapid cycling regimen of antiretroviral combination therapy in HIV-1 infected patients with virus harboring genotypic resistance to at least three classes of antiretroviral therapy.

The objectives are to study the feasibility, safety and efficacy of sequential combination therapy in HIV-1 infected patients with virus harboring genotypic resistance to at least three classes of antiretroviral agents and who currently have no adequate treatment options available.

This is an open-label, crossover, pilot study. Patients that fail their current regimen, and who currently have no adequate treatment options left, will be randomized to start either an alternating triple combination, or to start a continuous quadruple regimen of drugs. After 6 weeks, patients will crossover from either strategy to the other strategy for another 6 weeks. Each period is preceded by an interruption of all antiretroviral therapy for 4 weeks. In the study period when regimens are alternated, two combinations of three drugs with the least possible cross-resistance will alternate every week.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients
* At least 18 years of age
* Males or non-pregnant, non-lactating females
* Documented virological treatment failure on at least 3 classes of antiretroviral drugs
* No adequate antiretroviral therapy possible with currently available antiretroviral agents
* Virological treatment failure is defined as plasma HIV-1 RNA levels > 5000 while taking at least three different antiretroviral drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Changes in plasma HIV-1 RNA load | 12 weeks

SECONDARY OUTCOMES:
Changes in the genotype of the dominant quasispecies | 12 weeks
Replicative fitness of the dominant quasispecies | 12 weeks
Changes in CD4+ and CD8+ cell counts | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joep MA Lange, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Ferdinand Wit, MD PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- HIV Outpatient Clinic, Academic Medical Center, Amsterdam, North Holland, Netherlands